CLINICAL TRIAL: NCT05189782
Title: Mechanism of Resistance to GNC-038, a Tetra-specific T Cell Engager, in Relapsed and Refractory Diffuse Large B-cell Lymphoma
Brief Title: Mechanism of Resistance to GNC-038 in Relapsed and Refractory Diffuse Large B-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director of Shanghai Institute of Hematology, Ruijin Hospital
Other Study IDs: TRANS001-TeTE
Record Dates: First submitted 2021-09-03; First posted 2022-01-13 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects of the GNC-038 clinical trial (1): Patients enrolled in the GNC-038 Phase Ib/II clinical trial in Shanghai Ruijin Hospital.
- Non-malignant controls (2): Patients who have tonsillectomy due to obstructive sleep apnea and hyponea syndrome.

SUMMARY:
This is an exploratory study embedded in the Phase Ib/II clinical trial of CD3 x 4-1BB x CD19 x PD-L1 tetra-specific T cell engager GNC-038 in relapsed and refractory diffuse large B-cell lymphoma initiated by the corresponding pharmaceutical company. By measuring immune cell components and their functional phenotypes in peripheral blood and tumor tissues before and after the subject's medication, this study aims to identify key immune cell populations and immune molecules which play an important role in resistance to GNC-038 treatment, so as to optimize drug design and develop combination therapies to improve treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

For Group 1, the selection criteria are firstly concordant with those of the corresponding clinical trial. On this basis, additional selection criteria for this study are:

* Lymph node lesions with long diameter ≥ 2cm.
* Subjects have the ability and willingness to follow the visit, biosample collection and other research-related processes prescribed by the research program and to sign informed consent forms.

For Group 2, the selection criteria are:

* The subject is able to understand the informed consent form, and voluntarily participates and signs the informed consent form;
* Age between 18 and 80;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 points.

Exclusion Criteria:

For Group 1, the exclusion criteria are totally concordant with those of the corresponding clinical trial. There is no additional exclusion criteria for this study.

For Group 2, the exclusion criteria are:

* History of past or present malignant diseases;
* Patients with active autoimmune diseases, or patients with a history of autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's granulomatosis, polyvascular inflammation granuloma, Grave's disease, rheumatoid arthritis, pituitary inflammation, ophthalmic pigmentitis, autoimmune hepatitis, systemic sclerosis, Hashimoto thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain- Barre syndrome), etc.;
* Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection (HBsAg-positive or HBcAb-positive, HBV-DNA test positive), hepatitis C virus infection (HCV antibody-positive and HCV-RNA test positive), EB virus infection (EBV-DNA test positive), cytomegalovirus infection (CMV-DNA test positive) or herpes simplex virus infection (HSV-DNA test positive);
* Pregnant or nursing women;
* Previous organ transplants or allogeneic hematopoietic stem cell transplants;
* Under treatment of immunosuppressants, including but not limited to cyclosporine, tacrolimus, corticosteroids, etc., within 1 month prior to sampling;
* Fever (temperature >37.5 ℃) within 1 month prior to sampling, or using antibiotics due to respiratory, gastrointestinal, urinary tract infections, etc.;
* Other situations in which the researchers consider it inappropriate for the patient to participate in this study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study plans to include 10 subjects enrolled in the GNC-038 Phase Ib/II clinical trial in Ruijin Hospital. It also plans to include five patients who have tonsillectomy in Ruijin Hosptial due to obstructive sleep apnea and hyponea syndrome as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The abundance and phenotypes of immune cell subtypes within tumor or normal tonsil tissues measured by single-cell RNA sequencing. | In Group 1: change from screening to six weeks after treatment initiation, and to disease relapse or progression assessed up to 6 months after last treatment. In Group 2: immediately following tonsil resection.
  Core needle biopsies of lymph node lesions (in Group 1) or resected normal tonsil tissues (in Group 2) will be collected. 5' end single-cell RNA sequencing plus single-cell T cell receptor sequencing will be performed. The abundance and phenotypes of immune cell subtypes will be investigated using the above data.
The abundance and phenotypes of peripheral blood T cell subtypes measured by mass cytometry by the time-of-flight. | In Group 1: change from screening to day 22 and day 43 after treatment initiation, to 30 days after treatment ending, and to disease relapse or progression assessed up to 6 months after last treatment. In Group 2: within a week before tonsil resection.
  Peripheral blood mononuclear cells will be collected and mass cytometry by the time-of-flight will be performed to analyze a panel of T cell subtyping and functional surface molecules.

SECONDARY OUTCOMES:
Tumor cytogenetic and molecular genetic abnormalities. | During screening, six weeks after treatment initiation, and at disease relapse or progression assessed up to 6 months after last treatment.
  In Group 1, core needle biopsies of lymph node lesions will be collected, and whole exome sequencing will be performed to detect tumor cytogenetic and molecular genetic abnormalities. Peripheral blood mononuclear cells will also be collected and sequenced as healthy tissue reference.
Tumor gene expression profiles. | In Group 1: during screening, six weeks after treatment initiation, and at disease relapse or progression assessed up to 6 months after last treatment. In Group 2: immediately following tonsil resection.
  In Group 1, core needle biopsies of lymph node lesions will be collected, and bulk RNA sequencing will be performed to analyze gene expression profiles of tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China